CLINICAL TRIAL: NCT05003752
Title: Hypo-Combi Trial: Combined Hypofractionated External Beam Radiation Therapy (EBRT) Plus Interstitial High-Dose-Rate Brachytherapy (HDR-BT) Boost for Intermediate/High Risk Prostate Cancer
Brief Title: Hypo-Combi Trial: Hypofractionated EBRT Plus HDR-BT Boost for Prostate Cancer
Acronym: Hypo-Combi
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German Oncology Center, Cyprus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Not yet assigned
Record Dates: First submitted 2021-06-29; First posted 2021-08-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Prostate Adenocarcinoma; Radiation Toxicity
Keywords: HDR-Brachytherapy; EBRT; Prostate cancer
MeSH Terms: conditions — Radiation Injuries; Prostatic Neoplasms | interventions — Goserelin; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated EBRT plus HDR-BT boost (Other): Primarily hypofractionated EBRT consisting of 12 x 3 Gy/fraction, TD 36 Gy will be administered. Followed by HDR-BT boost of the prostate, TD 14 Gy.
  Interventions: Radiation: External beam radiation therapy, High-dose-rate brachytherapy; Drug: Goserelin 10.8 mg

INTERVENTIONS:
Radiation: External beam radiation therapy, High-dose-rate brachytherapy — Combined hypofractionated external beam radiation therapy (EBRT) plus high dose-rate brachytherapy (HDR-BT) schedule (total dose of EBRT 36 Gy/ in 12 fractions of 3 Gy plus HDR-BT with a total physical dose of 14 Gy in a single fraction)
Drug: Goserelin 10.8 mg — Androgen deprivation will be administered based on NCCN guidelines in patients with unfavorable intermediate/high risk organ-confined prostate cancer
  Other Names: Androgen deprivation therapy (upon indication)

SUMMARY:
Hypo-Combi Trial: A Prospective Phase I/II Study of Combined Hypofractionated External Beam Radiation Therapy (EBRT) plus Interstitial High-Dose-Rate Brachytherapy (HDR-BT) for Intermediate/High Risk Prostate Cancer

DETAILED DESCRIPTION:
The Phase I/II trial will prospectively assess the acute, early late and late gastrointestinal (GI), genitourinary (GU) and sexual toxicity of combined hypofractionated external beam radiation therapy (EBRT) plus high dose-rate brachytherapy (HDR-BT) schedule (total dose of EBRT 36 Gy/ in 12 fractions of 3 Gy plus HDR-BT with a total physical dose of 14 Gy in a single fraction) for patients with unfavourable intermediate/high risk (based on NCCN stratification guidelines) organ-confined prostate cancer, not requiring pelvic irradiation.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form
* Age > 18 years old.
* Life expectancy of at least five years, excluding his diagnosis of prostate cancer.
* Histopathologically proven primary adenocarcinoma of the prostate
* The patient must be registered within 180 days following the histopathological confirmation of the malignancy
* Prostate volume < 80ml
* International Prostate Symptom Score (IPSS) < 18
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients with a history of non-prostate malignancies are eligible if they have been disease-free for 5 or more years prior to enrolment, are deemed by their physician to be at low risk for recurrence and they did not need pelvic radiotherapy as part of their treatment. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria:

* Histopathological confirmation or suspicion in conventional or molecular imaging of regional or distant metastases
* Prior pelvic radiotherapy
* Known autoimmune disorders (e.g. inflammatory bowel disease, lupus, scleroderma)
* Prior TURP
* MRI non compatible metal implants
* Pre-existing fistulae
* Contraindication for general and spinal anaesthesia
* Inability to be placed in lithotomy position
* Any treatment with radiation therapy, chemotherapy, immunotherapy, biotherapy and/or hormonal therapy for the currently diagnosed prostate cancer prior to registration.
* History of non-prostate malignancy, apart from patients that have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of acute and early late genitourinary, gastrointestinal and sexual toxicity | up to 2 years
  RTOG/EORTC questionnaires will be collected and evaluated for GU/GI toxicity. International Prostate Symptom Score will be assessed for lower urinary tract symptomatology and IIEF-5 for erectile function.

SECONDARY OUTCOMES:
Rate of biochemical control | 2 years, 5 years
  Evaluation of 2- and 5-year biochemical control based on the Phoenix criteria
Rate of overall survival | 2 years, 5 years
  Evaluation of 2- and 5-year overall survival rate
Rate of prostate cancer-specific survival | 2 years, 5 years
  Evaluation of 2- and 5-year prostate cancer-specific survival rate
Rate of distant metastasis-free survival | 2 years, 5 years
  Evaluation of 2- and 5-year distant metastasis-survival rate
Rate of treatment-related symptoms on Quality of Life assessed by Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) questionnaire | 2 years, 5 years
  Record quality of life (QOL) issues related to treatment-related symptoms and overall satisfaction. Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) questionnaire will be used. Minimum score is 0 points and maximum score is 60 points, with lower points meaning better quality of life and higher point score meaning, alternatively, worse outcome.
18F-PSMA PET/CT Vs conventional imaging for identification of pelvic nodal or distant secondaries | 2 years
  Evaluation of the accuracy of first-line imaging for identifying either pelvic nodal or distant-metastatic disease defined by the receiver-operating curve using a predefined reference-standard including histopathology, imaging, and biochemistry at 6-month follow-up and compare to 18F-PSMA PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Strouthos, MD PhD, Principal Investigator — German Oncology Center, Cyprus
Locations (1):
- German Oncology Center, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No
Data regarding this study will be presented at international meetings. Manuscripts will be submitted to peer-reviewed Journals